CLINICAL TRIAL: NCT04895826
Title: Computer-vision Aided Community Back Pain Physiotherapy Services
Acronym: CV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oxford Brookes University (Other)
Collaborators: Good Boost Wellbeing (Unknown); National Axial Spondyloarthritis Society (Unknown)
Responsible Party: Principal Investigator, Helen Dawes, Professor, Oxford Brookes University
Other Study IDs: 201429
Record Dates: First submitted 2021-05-15; First posted 2021-05-20 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Back Pain; Healthy Control
Keywords: Posture Movement Back pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Back pain and no back pain: Participants with and without back pain will be included in the study and they will be asked to perform standard functional movements that would be used for a physiotherapy assessment for a back condition. The participants will also perform these movements in front of a camera for video recordings to be analysed by the CV system. The measurements by the CV system will be compared to the measurements by the physiotherapist. Additionally, participants will perform and record videos of the same set of movements at home to test the feasibility of the CV system in a home environment.

SUMMARY:
Back pain affects one-third of the UK population every year with a huge impact on the health service and economy. The aim of this study is to test the validity of a computer-vision (CV) technology that uses cameras on phones/tablets/webcams to assess a person's movement and function with the ultimate goal to use the CV system to screen for back pain conditions. Participants with and without back pain will be included in the study and they will be asked to perform standard functional movements that would be used for a physiotherapy assessment for a back condition. The participants will also perform these movements in front of a camera for video recordings to be analysed by the CV system. The measurements by the CV system will be compared to the measurements by the physiotherapist. Additionally, participants will perform and record videos of the same set of movements at home to test the feasibility of the CV system in a home environment.

DETAILED DESCRIPTION:
Back pain affects one-third of the UK population every year with a huge impact on the health service and economy. One specific back pain condition is Axial Spondyloarthropathy (AxSpa), which is an inflammatory spinal arthritis that causes pain and stiffness. This life-long condition presents in the early twenties as 'regular' back pain. Due to its similarity to other back pain conditions, there is an average 8.5-year delay to diagnosis. The aim of this study is to test the validity of a computer-vision (CV) technology that uses cameras on phones/tablets/webcams to assess a person's movement and function with the ultimate goal to use the CV system to screen for back pain conditions, such as AxSpa. The CV system development is led by the GoodBoost Wellbeing Limited and The National Axial Spondyloarthritis Society (NASS) is supporting the recruitment of people living with AxSpa.

The CV system that has been developed is a form of artificial intelligence video analysis which is able to automatically measure specific functional movements captured on video. To validate this CV system, this study is designed to compare it to the clinical gold standard measurement by a physiotherapist. Participants with and without back pain will be included in the study and they will be asked to perform standard functional movements that would be used for a physiotherapy assessment for a back condition. The participants will also perform these movements in front of a camera for video recordings to be analysed by the CV system. The measurements by the CV system will be compared to the measurements by the physiotherapist. Additionally, participants will perform and record videos of the same set of movements at home to test the feasibility of the CV system in a home environment.

ELIGIBILITY:
Inclusion Criteria:

* ● The participant is willing and able to give informed consent for participation in the study.

  * Male or Female, aged 18 years or above.
  * For back pain group: diagnosed with AxSpa or long-standing non-specific LBP
  * For healthy group: healthy with no long-standing back pain
  * For the home setting, the participant must be capable of uploading videos from a smartphone or webcam.

Exclusion Criteria:

* ● Has had surgery within 6 months of registration

  * Unable to stand independently
  * Unable to pass screening questions to participate in physical activity
  * Serious neurological condition preventing normal movement or walking ability
  * Any severe medical conditions, such as cardiovascular disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy participants and participants with non-specific back pain will be recruited via advertisement through networks associated with the research team members. Participants with AxSpa will initially be recruited from the Oxford area by The National Axial Spondyloarthritis Society (NASS) promotion.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Primary movement Lumbar spine lateral flexion | 1 minute
  Concurrent validity of lumbar spine lateral flexion measurement by the CV system compared to physiotherapy measurement.

SECONDARY OUTCOMES:
Movement of Lumbar global flexion | 1 minute
  Concurrent validity of: Lumbar global flexion measurement by the CV system compared to physiotherapy measurement.
Movement of Cervical rotation | 1 minute
  Concurrent validity of: Cervical rotation seated measurement by the CV system compared to physiotherapy measurement.
Movement of Hip internal rotation | 1 minute
  Concurrent validity of: Hip internal rotation seated measurement by the CV system compared to physiotherapy measurement.
Movement of Hip abduction | 1 minute
  Concurrent validity of: Hip abduction standing measurement by the CV system compared to physiotherapy measurement.
Movement of Shoulder flexion | 1 minute
  Concurrent validity of: Shoulder flexion measurement by the CV system compared to physiotherapy measurement.
Movement 6 | 1 minute
  Concurrent validity of: Chest expansion measurement by the CV system compared to physiotherapy measurement.
Movement of Sit-to-stand | 1 minute
  Concurrent validity of Sit-to-stand measurement by the CV system compared to physiotherapy measurement.
Standing posture spinal kyphosis | 1 minute
  Posture as measured by spinal kyphosis
Standing posture tragus to ear | 1 minute
  Posture as measured by tragus to walk
Leg strength | 1 minute
  5 time sit to stand

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Brookes, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Direct access will be granted to authorised representatives from the Sponsor and host institution for monitoring and/or audit of the study to ensure compliance with regulations.